CLINICAL TRIAL: NCT03564067
Title: Maintaining Response With tDCS in Depression (MARt- Depression) Pilot Study
Brief Title: MARt-Depression Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Chair, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 126-2016
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Major Depressive Disorder
Keywords: TRD; tDCS; cCBT; Home-based tDCS-cCBT
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS + cCBT (Other): After baseline assessments are complete, participants will be provided with a tDCS device (Soterix Medical tDCS mini-Clinical Trials system (mini-CT)), which is deactivated until a code is provided by the research staff. Each tDCS session will be delivered in combination with a computerized CBT module and participants will progress through the computerized CBT course (Beacon Therapist-Assisted-Internet-Delivered CBT) over the 6 months of treatment at their own pace.
  Interventions: Device: Soterix Medical tDCS mini-Clinical Trials system (mini-CT); Behavioral: Computerized CBT (cCBT)

INTERVENTIONS:
Device: Soterix Medical tDCS mini-Clinical Trials system (mini-CT) — Participants are provided with an activation code. This code will unlock a single session with the pre-set 30 minute duration and intensity (direct current 2mA, current density 0.80A/m2, with anode over the left and cathode over the right dorsolateral prefrontal cortex, respectively). Home-based tDCS will involve 30-min tDCS (3 days per week) for the first 3 months and once weekly for the subsequent 3 months.
Behavioral: Computerized CBT (cCBT) — Each tDCS session will be delivered in combination with a computerized CBT module and participants will progress through the computerized CBT course (Beacon Therapist-Assisted-Internet-Delivered CBT) over the 6 months of treatment at their own pace.

SUMMARY:
This is an open label pilot feasibility study that will recruit 15 participants. The purpose of the pilot study will be to evaluate the feasibility of open label Transcranial direct current stimulation (tDCS) in combination with computerized cognitive behavior therapy (cCBT) to maintain wellness following an acute course of Electroconvulsive therapy (ECT) for up to 6 months.

DETAILED DESCRIPTION:
Home-based tDCS-cCBT will involve 30-min tDCS (3 days per week) for the first 3 months and once weekly for the subsequent 3 months, in combination with computerized CBT delivered through an online portal for the duration of tDCS each day. Subjects who miss 4 consecutive treatment days or 20 percent of total treatments will be excluded from the study as it is our intention to encourage compliance with the proposed treatments to maintain optimal wellness. All missed treatment days will be recorded in a log for each participant.

Aim 1. To investigate the effectiveness of maintenance tDCS-cCBT for patients with MDD who have responded to a successful acute course of ECT.

Hypothesis 1. tDCS-cCBT will effectively maintain treatment response in MDD in a manner that is non-inferior to that of maintenance ECT.

ELIGIBILITY:
Inclusion Criteria:

1. History of Major Depressive Disorder with most recent episode treated with acute ECT at the Temerty Centre for Therapeutic Brain Intervention, CAMH.
2. Individuals capable to provide consent who are receiving care as outpatients, and are now remitters (defined by the 24-item Hamilton Rating Scale for Depression (HRSD-24) ≤ 10).
3. Age 18-85, inclusive.

Exclusion Criteria:

1. History of a DSM-IV substance use disorder within the past three months
2. Concomitant major unstable medical illness
3. Pregnancy or the intention to become pregnant during the study
4. DSM-IV diagnosis of any psychotic disorder, obsessive compulsive disorder, or post-traumatic stress disorder (current or within the last year) as confirmed by the Mini-International Neuropsychiatric Interview (MINI)
5. DSM-IV diagnosis of personality disorder as assessed by a study investigator
6. Baseline score of < 24 on the MoCA
7. Any significant neurological disorder (e.g., a space occupying brain lesion, a history of stroke, a cerebral aneurysm, a seizure disorder, Parkinson's disease, Huntington's chorea, multiple sclerosis, head trauma with loss of consciousness for greater than or equal to five minutes)
8. Presenting with a medical condition, a medication, or a laboratory abnormality that could cause a major depressive episode or significant cognitive impairment in the opinion of the investigator (e.g., hypothyroidism with low TSH, Cushing's disease)
9. Any intracranial implant (e.g., aneurysm clips, shunts, cochlear implants) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
10. Any dermatological disorder or any cuts/broken skin in the scalp region that may affect the safe delivery of the tDCS stimulus
11. Requiring a benzodiazepine with a dose equivalent to lorazepam 2 mg/day or higher or any anticonvulsant due to the potential of these medications to limit the efficacy of ECT
12. The inability to communicate in spoken and written English fluently enough to complete the neuropsychological tests due to a language barrier or a non-correctable clinically significant sensory impairment (i.e., cannot hear or see well enough to complete the neuropsychological tests).
13. Cognitive impairment or physical impairment such that they are unable to learn to, or physically unable to apply tDCS to their scalp without assistance (after training).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-07-05 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Maintained remission of depressive symptoms as measured by the Hamilton Rating Scale for Depression - 24 | 6 months
  Hamilton Rating Scale for Depression (24-item version)
  * This scale is used to quantify the severity of symptoms of depression
  * Scale range: 0-76 (total score)
  * Lower scores indicate lower severity of depressive symptoms (i.e., better outcome)
  * Higher scores indicate higher severity of depressive symptoms (i.e., worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Zafiris J Daskalakis, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital — http://www.camh.net/research